CLINICAL TRIAL: NCT03116620
Title: Chewing Function in Pediatric Neuromuscular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Chewing in pediatric NMD
Record Dates: First submitted 2017-04-11; First posted 2017-04-17 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Mastication Disorder
Keywords: mastication; children with neuromuscular disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chewing evaluation (Experimental): Children with neuromuscular disorders (NMD) will be participated. Children will be asked to chew a standardized biscuit while video recording. Two physical therapists will assess all video recordings independently and score each video according to the KCPS. The correlation between the KCPS scores of two therapists will be used for interobserver reliability. One therapist will rescore the recordings after an interval of 2 weeks for intraobserver reliability.
  Interventions: Other: Chewing evaluation

INTERVENTIONS:
Other: Chewing evaluation — Children with neuromuscular disorders (NMD) will be participated. Children will be asked to chew a standardized biscuit while video recording. Two physical therapists will assess all video recordings independently and score each video according to the KCPS. The correlation between the KCPS scores of two therapists will be used for interobserver reliability. One therapist will rescore the recordings after an interval of 2 weeks for intraobserver reliability.

SUMMARY:
We aimed to evaluate chewing function (CF) in children with neuromuscular disorders, and investigate reliability of the Karaduman Chewing Performance Scale (KCPS).

DETAILED DESCRIPTION:
Chewing disorders (CD) can be seen due to muscle weakness in children with neuromuscular disorders neuromuscular disorders (NMD). Normal diet consists of all food consistencies including liquid, pudding and solid foods, and CD causes inability to intake solid food. This condition can affect development, nutritional behavior and child-parent interaction in children. Thus, it is important to determine CD in an early period with appropriate assessment methods and plan appropriate therapies in NMD. We aimed to evaluate chewing function (CF) in children with NMD, and investigate reliability of the Karaduman Chewing Performance Scale (KCPS).

ELIGIBILITY:
Inclusion Criteria:

* Children above the age of 2 years
* Children with neuromuscular disorders

Exclusion Criteria:

* Children under the age of 2 years
* Children without neuromuscular disorders

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
The reliability of the KCPS in children with neuromuscular disorders | 1 month
  Children with neuromuscular disorders (NMD) will be participated. Children will be asked to chew a standardized biscuit while video recording. Two physical therapists will assess all video recordings independently and score each video according to the KCPS. The correlation between the KCPS scores of two therapists will be used for interobserver reliability. One therapist will rescore the recordings after an interval of 2 weeks for intraobserver reliability.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No